CLINICAL TRIAL: NCT01686568
Title: Dietary Omega-3 Fatty Acids as a Therapeutic Strategy in Insulin Resistant Humans
Brief Title: Omega-3 Fatty Acids and Insulin Sensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Building Interdisciplinary Research Careers in Women's Health (Unknown)
Responsible Party: Principal Investigator, Ian R. Lanza, Assistant Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-004590; KL2TR000136 (NIH); U24DK100469 (NIH); DK50456 (Other Grant/Funding Number: Minnesota Obesity Center); DK40484 (Other Grant/Funding Number: Minnesota Obesity Center); 5T32DK007352 (NIH); 5UL1TR000135 (NIH)
Record Dates: First submitted 2012-09-11; First posted 2012-09-18 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Docosahexaenoic Acids; Fatty Acids, Essential; Fatty Acids, Omega-3; Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omega-3 (Experimental): Patients in this group will receive oral supplementation with EPA+DHA (3.9grams/day) for 6 months.
  Interventions: Drug: Omega-3
- Placebo (Placebo Comparator): Patients in this group will be supplemented with placebo capsules containing ethyl oleate.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Omega-3 — Patients in this group will receive oral supplementation with EPA+DHA (3.9grams/day) for 6 months.
  Other Names: Essential fatty acids; Omega-3 fatty acids; Omega-3 polyunsaturated fatty acids; PUFAs; Lovaza
  Arms: Omega-3
Drug: placebo
  Arms: Placebo

SUMMARY:
This study is being done to understand the effects of dietary omega-3 fats on insulin sensitivity in adult men and women.

DETAILED DESCRIPTION:
Dietary omega-3 polyunsaturated fatty acids (n-3 PUFA), which include eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) from fish oil, prevent insulin resistance in rodents, but data in humans is ambiguous. No existing studies have systematically evaluated the influence of n-3 PUFAs on insulin sensitivity and beta cell function in insulin resistant, non-diabetic humans. The Investigators hypothesize that 6 months of oral supplementation of purified EPA/DHA (3.9g/day) will significantly improve hepatic and peripheral insulin sensitivity and beta cell responsiveness in insulin-resistant, non-diabetic individuals. Based on recent work in mice, the investigators also hypothesize that EPA/DHA will increase the content and function of mitochondria in skeletal muscle, measured using a combination of in vivo and in vitro methods. Overall, the investigators hypothesize that EPA+DHA supplementation will improve hepatic and peripheral insulin sensitivity in insulin resistant humans, and this improvement will be associated with mitochondrial biogenesis and attenuated lipid accumulation in skeletal muscle and liver.

A sub-study was added in which participants receiving dietary omega-3 fatty acids or placebo supplements underwent abdominal subcutaneous adipose tissue biopsies to measure the content of total, pro- (M1) and anti- (M2) inflammatory macrophages (immunohistochemistry), crown-like structures (immunohistochemistry), and senescent cells (β-galactosidase staining), as well as a two-step euglycemic, pancreatic clamp with a stable-isotope labeled precursor ((U-13C)palmitate) infusion to determine the insulin concentration needed to suppress palmitate flux by 50% (IC50(palmitate)f).

ELIGIBILITY:
Inclusion criteria:

1. Age 18-65 years
2. Insulin resistant (Homeostasis Model Assessment (HOMA) Insulin Resistance (IR) ≥2.6)

Exclusion criteria:

1. Current use of omega-3 nutritional supplements
2. Fasting plasma glucose ≥126 mg/dL
3. Active coronary artery disease
4. Participation in structured exercise (>2 times per week for 30 minutes or longer)
5. Smoking
6. Medications known to affect muscle metabolism (e.g., beta blockers, corticosteroids, tricyclic-antidepressants, benzodiazepines, opiates, barbiturates, anticoagulants)
7. Renal failure (serum creatinine > 1.5mg/dl)
8. Chronic active liver disease (AST>144 IU/L and alanine transaminase (ALT)>165 IU/L)
9. Anti-coagulant therapy (warfarin/heparin)
10. International normalized ratio (INR) >3
11. Use of systemic glucocorticoids
12. Chronic use of NSAIDS or aspirin
13. Pregnancy or breastfeeding
14. Alcohol consumption greater than 2 glasses/day
15. Hypothyroidism
16. Fish or shellfish allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-12-21 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2015-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Lanza, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Lalia AZ, Johnson ML, Jensen MD, Hames KC, Port JD, Lanza IR. Effects of Dietary n-3 Fatty Acids on Hepatic and Peripheral Insulin Sensitivity in Insulin-Resistant Humans. Diabetes Care. 2015 Jul;38(7):1228-37. doi: 10.2337/dc14-3101. Epub 2015 Apr 7. PMID 25852206
- [Derived] Hames KC, Morgan-Bathke M, Harteneck DA, Zhou L, Port JD, Lanza IR, Jensen MD. Very-long-chain omega-3 fatty acid supplements and adipose tissue functions: a randomized controlled trial. Am J Clin Nutr. 2017 Jun;105(6):1552-1558. doi: 10.3945/ajcn.116.148114. Epub 2017 Apr 19. PMID 28424185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Mayo Clinic in Rochester, Minnesota.
Groups:
- Omega-3: Patients in this group will receive oral supplementation with EPA + Docosahexaenoic acid (DHA) (3.9grams/day) for 6 months.
Period: Main Study
Arm/Group | Omega-3 | Placebo
Started | 16 | 15
Completed | 14 | 11
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Noncompliance with protocol | 0 | 1
Not completed — Liver enzymes above range of exclusion | 1 | 0
Period: Sub-Study
Arm/Group | Omega-3 | Placebo
Started | 14 | 11
Completed | 12 | 9
Not Completed | 2 | 2
Not completed — Not consented for sub-study | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for participants who received treatment and did not withdraw from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 | Placebo | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (2.9) | 32.6 (2.5) | 34.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity by Hyperinsulinemic-euglycemic Clamp at Baseline and 6 Month Follow up
Description: A 2-stage insulin clamp will be performed with titration of dextrose to maintain euglycemia. D2 glucose will be infused to evaluate hepatic glucose production at baseline and in response to insulin. Hyperinsulinemic-euglycemic clamp technique: The plasma insulin concentration is acutely raised and maintained by a continuous infusion of insulin. Meanwhile, the plasma glucose concentration is held constant at basal levels by a variable glucose infusion. When the steady-state is achieved, the glucose infusion rate (GIR) equals glucose uptake by all the tissues in the body and is therefore a measure of tissue insulin sensitivity.
Time Frame: Baseline, after 6 months of treatment
Measure: Mean (Standard Error); unit: mg/kg FFM/min
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 14 | 11
mg/kg FFM/min
  Baseline | 10.92 (1.04) | 10.39 (0.76)
  6 Month Follow Up | 10.16 (1.02) | 10.80 (0.73)

2. Secondary Outcome: Beta Cell Function From Insulin Secretion Following Ingestion of a Mixed Meal at Baseline and 6 Month Follow up
Description: Following consumption of a mixed meal, beta cell function will be evaluated from serial measurements of C-peptide. C-peptide was measured using a two-side immunometric assay using electrochemiluminescence detection.
Time Frame: baseline, after 6 months of treatment
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 14 | 11
nmol/L
  Baseline | 537.17 (45.33) | 488.90 (45.47)
  6 Month Follow Up | 561.33 (48.21) | 504.39 (35.93)

3. Secondary Outcome: Mitochondrial Function Determined by Muscle Biopsy at Baseline and 6 Month Follow up
Description: Measurements of oxygen consumption in isolated mitochondria will be performed using a polarographic oxygen electrode.
Time Frame: Baseline, after 6 months of treatment
Measure: Mean (Standard Error); unit: pmol/s/mg tissue
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 14 | 11
pmol/s/mg tissue
  Baseline | 496.81 (26.54) | 564.86 (42.10)
  6 Month Follow Up | 406.38 (40.39) | 495.12 (39.79)

4. Secondary Outcome: Insulin Concentration Needed to Suppress Palmitate Appearance Rates (IC50(Palmitate)f)
Description: Sensitivity of adipose tissue lipolysis to insulin suppression, was calculated as the insulin concentration needed to suppress palmitate appearance rates (ie, flux) by 50% (IC50(palmitate)f).
Time Frame: approximately after 6 months of treatment
Population: The number of subjects analyzed for this outcome measure for the placebo arm was 8 instead of 9. One subject did not have blood drawn for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: µU/mL
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 12 | 8
µU/mL
  Baseline | 22 [13 to 24] | 25 [22 to 33]
  Post-intervention | 18 [16 to 29] | 19 [14 to 46]

5. Secondary Outcome: Senescent Cells
Description: Tissue burden of senescent cells, which was measured by staining for senescence-associated B-galactosidase activity and expressed as the number per 100 nucleated positive cells.
Time Frame: approximately after 6 months of treatment
Measure: Mean (Standard Deviation); unit: number positive cells/100 total cells
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 12 | 9
number positive cells/100 total cells
  Baseline | 4 (3) | 4 (3)
  Post-intervention | 4 (3) | 4 (2)

6. Secondary Outcome: Immunohistochemistry Assessments of Macrophage Burden
Description: One week after the pancreatic clamp study, participants were provided a standardized meal before an overnight fast. The next morning an abdominal adipose tissue biopsy was collected, and the samples were analyzed for adipocyte size. Immunohistochemistry was used to assess macrophage burden (total (CD68), M1 (CD14) and M2 (CD206) macrophages per 100 adipocytes).
Time Frame: approximately after 6 months of treatment
Measure: Mean (Standard Deviation); unit: macrophages per 100 adipocytes
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 12 | 9
macrophages per 100 adipocytes
  Total (CD68) baseline | 31 (8) | 33 (5)
  Total (CD68) post intervention | 33 (8) | 31 (5)
  M1 (CD14) baseline | 11 (6) | 13 (4)
  M1 (CD14) post intervention | 14 (6) | 12 (5)
  M2 (CD206) baseline | 28 (5) | 29 (7)
  M2 (CD206) post intervention | 29 (9) | 29 (5)

7. Secondary Outcome: Macrophage Crown-like Structures
Description: Macrophages surrounding dying or dead adipocytes form crown-like structures (CLSs). One week after the pancreatic clamp study, participants were provided a standardized meal before an overnight fast. The next morning an abdominal adipose tissue biopsy was collected, and the samples were analyzed for adipocyte size. Immunohistochemistry was used to assess the number of crown-like structures per 10 images.
Time Frame: approximately after 6 months of treatment
Measure: Median (Inter-Quartile Range); unit: crown-like structures per 10 images
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 12 | 9
crown-like structures per 10 images
  Baseline | 0 [0 to 1] | 1 [0 to 3]
  Post-intervention | 0 [0 to 1] | 1 [0 to 2]

8. Post Hoc Outcome: EPA and DHA Concentrations in Plasma
Description: Post hoc analyses were conducted to test whether EPA and DHA concentrations in plasma in response to intervention explained variation in outcome measures of adipose tissue lipolysis insulin sensitivity and inflammatory markers post-intervention.
Time Frame: approximately after 6 months of treatment
Measure: Mean (Standard Error); unit: percentage of total free fatty acid
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 12 | 9
percentage of total free fatty acid
  EPA Baseline | 0.95 (0.22) | 1.2 (0.27)
  EPA Post-Intervention | 6.0 (0.92) | 1.1 (0.19)
  DHA Baseline | 0.89 (0.23) | 1.2 (0.39)
  DHA Post-Intervention | 3.5 (0.84) | 0.90 (0.18)

9. Post Hoc Outcome: EPA and DHA Concentrations in Adipose Tissue
Description: Post hoc analyses were conducted to test whether EPA and DHA concentrations in subcutaneous abdominal adipose tissue in response to intervention explained variation in outcome measures of adipose tissue lipolysis insulin sensitivity and inflammatory markers post-intervention.
Time Frame: approximately after 6 months of treatment
Measure: Mean (Standard Error); unit: percentage of total free fatty acid
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 12 | 9
percentage of total free fatty acid
  EPA baseline | 0.06 (0.00) | 0.07 (0.01)
  EPA Post-Intervention | 0.19 (0.02) | 0.07 (0.01)
  DHA Baseline | 0.14 (0.01) | 0.15 (0.01)
  DHA Post-Intervention | 0.28 (0.02) | 0.16 (0.02)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Omega-3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes